CLINICAL TRIAL: NCT04092400
Title: Prospective Observational Study of Patients Implanted With Micro-invasive Glaucoma Surgical (MIGS) Devices at the National University Hospital, Singapore
Brief Title: Study on Micro-invasive Glaucoma Surgical (MIGS) Devices
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: DSRB - 2016/00125
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-09

CONDITIONS: Glaucoma
Keywords: Glaucoma; Glaucoma Surgery; Minimally Invasive Surgery
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Micro-Invasive Glaucoma Surgical devices: Patients implanted With Micro-invasive Glaucoma Surgical (MIGS) devices at the National University Hospital, Singapore
  Interventions: Device: Micro-invasive Glaucoma Surgical Devices

INTERVENTIONS:
Device: Micro-invasive Glaucoma Surgical Devices — Safety and efficacy of Micro-invasive Glaucoma Surgical Devices

SUMMARY:
Glaucoma is an ocular condition in which optic nerve damage occurs, frequently in the presence of increased pressure within the eye. Micro-invasive glaucoma surgery (MIGS) refers to a new group of surgical procedures which are characterized by the following features: high safety profile, minimal trauma, ease of use and rapid recovery. There are 3 main groups of MIGS devices, which drain fluid to different regions in the eye: the Schlemm's canal, the suprachoroidal space and the subconjunctival space. Though MIGS devices were introduced in the United States of America, Canada and Europe more than 5 years ago, and have attained the CE mark and FDA approval for some devices. Studies have shown that these devices have a high safety profile and are effective (1-5). However, MIGS devices are only recently available in Asia, and data on their clinical outcomes in Asian patients are limited.

DETAILED DESCRIPTION:
* Data will be collected for 5 years after surgery, and the data collected will be the routine examination findings and investigations before and after surgery (as part of standard medical treatment)
* Visual acuity testing, refraction, humphrey perimetry, heidelberg retinal tomography, anterior segment optical coherence tomography, pre-operative endothelial cell count, corneal pachymetry, intraocular pressure measurement, number of glaucoma medications
* A log will be used to keep track of subject's wishes on the return for incidental findings (IF) according to subject's choice during the signing of consent form (however, we do not anticipate any incidental findings related to the study as this is an observational and non-interventional study).
* In case of return incidental finding for subject who consented, PI will inform the research subject, or his legally authorised representatives, information and feedback on IFs.
* PI with sufficient time for explanation and for the research subject to ask questions.
* Sufficient information will be provided to the research subject or his legally authorised representative so that he can make an informed decision as to whether to return to the Institution for medical consultation, seek an opinion elsewhere, or to have no follow-up action with regards to the IF.

Sample size and power calculations are not applicable as this observational study involves Medical Records Review and is not an interventional study.The recruitment target of 500 is based on the upper limit of the estimated number of patients who will undergo micro-invasive glaucoma surgical device implantation during the study period, though it is likely to be an overestimation. Pre-operative intraocular pressure and number of glaucoma medications will be compared with post-operative intraocular pressure and number of glaucoma medications at one year, 2 years, 3 years, 4 years and 5 years after surgery, using the paired t-test. Statistical significance is set at p<0.05

All activities involving the patient will be performed as part of the routine diagnostic or standard medical treatment as part of the subject's standard care. This is an observational study and no activities outside standard care will be performed as part of this study.The activities not involving the patient includes screening, data collection, data analysis.

ELIGIBILITY:
Inclusion Criteria:

* are all patients with glaucoma who have been listed for implantation of micro-invasive glaucoma surgical devices, with or without cataract surgery

Exclusion Criteria:

* Advanced glaucoma (as defined as cup-disc ratio ≥ 0.9 and/or a visual field defect within central 10˚ of fixation) ; diagnosis of glaucoma other than POAG and PACG (including uveitic, neovascular, traumatic glaucoma or glaucoma secondary to raised episcleral venous pressure); prior incisional glaucoma surgery or cataract surgery; presence of scarring, prior surgery or other conjunctival pathologies in the target quadrant; presence of vitreous in the anterior chamber; presence of intraocular silicone oil; clinically significant inflammation or infection in the study eye within 30 days before the pre-operative visit; known or suspected allergy or sensitivity to drugs required for the surgery (including anaesthesia) or any of the device components (eg. porcine products and glutaraldehyde); and any corneal, choroidal, retinal, orbital disease which may interfere with MIGS device implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Glaucoma patients undergoing micro-invasive glaucoma surgical devices, with or without cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-03-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) reduction | 12 months
  IOP reduction at 12 months compared with baseline unmedicated IOP

SECONDARY OUTCOMES:
Reduction in topical glaucoma medication | 12 months
  Topical glaucoma medication use at 12 months, the incidence of complications and failure

CONTACTS AND LOCATIONS:
Overall Officials: Chelvin Sng, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Chelvin Sng, National University Hospital Department of Ophthalmology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD

REFERENCES:
- [Background] Garcia-Feijoo J, Rau M, Grisanti S, Grisanti S, Hoh H, Erb C, Guguchkova P, Ahmed I, Grabner G, Reitsamer H, Shaarawy T, Ianchulev T. Supraciliary Micro-stent Implantation for Open-Angle Glaucoma Failing Topical Therapy: 1-Year Results of a Multicenter Study. Am J Ophthalmol. 2015 Jun;159(6):1075-1081.e1. doi: 10.1016/j.ajo.2015.02.018. Epub 2015 Mar 3. PMID 25747677
- [Result] Hengerer FH, Auffarth GU, Riffel C, Conrad-Hengerer I. Second-Generation Trabecular Micro-Bypass Stents as Standalone Treatment for Glaucoma: A 36-Month Prospective Study. Adv Ther. 2019 Jul;36(7):1606-1617. doi: 10.1007/s12325-019-00984-9. Epub 2019 May 22. PMID 31119690
- [Result] Saheb H, Ahmed II. Micro-invasive glaucoma surgery: current perspectives and future directions. Curr Opin Ophthalmol. 2012 Mar;23(2):96-104. doi: 10.1097/ICU.0b013e32834ff1e7. PMID 22249233
- [Result] Shah M, Law G, Ahmed II. Glaucoma and cataract surgery: two roads merging into one. Curr Opin Ophthalmol. 2016 Jan;27(1):51-7. doi: 10.1097/ICU.0000000000000224. PMID 26569527
- [Result] Ahmed II. MIGS and the FDA: What's in a Name? Ophthalmology. 2015 Sep;122(9):1737-9. doi: 10.1016/j.ophtha.2015.06.022. No abstract available. PMID 26299720